CLINICAL TRIAL: NCT05797623
Title: A Multicenter, Randomized, Double-blind, and Open-label, Placebo-controlled Phase II Clinical Study of Trappa Ethanolamine Tablets Combined With Ciclosporin in Patients With Treatment of Non-severe Aplastic Anemia
Brief Title: Safety and Effectiveness of Trappa Ethanolamine Tablets Combined With Ciclosporin in the Treatment of Primary Treatment of Non-severe Aplastic Anemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR8735-201
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-03

CONDITIONS: Non-severe Aplastic Anemia
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trappa ethanolamine tablets combined with ciclosporin (Experimental)
  Interventions: Drug: Trappa ethanolamine tablets ; ciclosporin
- Placebo combined with ciclosporin (Placebo Comparator)
  Interventions: Drug: Placebo ; ciclosporin

INTERVENTIONS:
Drug: Trappa ethanolamine tablets ; ciclosporin — Trappa ethanolamine tablets combined with ciclosporin
  Arms: Trappa ethanolamine tablets combined with ciclosporin
Drug: Placebo ; ciclosporin — Placebo combined with ciclosporin
  Arms: Placebo combined with ciclosporin

SUMMARY:
This is a multicenter, randomized, double-blind, and open-label, placebo-controlled phase II clinical study. In order to evaluate the effectiveness and safety of trappa ethanolamine tablets combined with ciclosporin in the treatment of patients with non-severe aplastic anemia.

ELIGIBILITY:
Inclusion Criteria:

1. 14-75 years old (including boundary value, whichever is at the time of signing the informed consent form), Gender is not limited.
2. Diagnosed with non-heavy aplastic anemia within 6 months
3. Life Functional Status (ECOG) Score 0-1
4. Those who understand the research procedures and methods, voluntarily participate in this experiment, and sign the informed consent form in writing

Exclusion Criteria:

1. Total blood cell loss and myelohypoproliferative diseases caused by other reasons
2. Chromosome karyotype analysis during screening shows clonal cytogenetic abnormalities
3. Meet the severe aplastic anemia
4. Paroxysmal sleep hemoglobinuria (PNH) clone ≥50% or hemolytic PNH clone
5. Randomly receive ATG, ciclosporin, TPO-R agonists, androgens and other drugs to treat the relapse without completing the elution
6. Pre-randomized treatment with erythropoietin
7. Pre-randomized use of corticosteroids, G-CSF and GM-CSF treatment
8. People with a history of hematopoietic stem cell transplantation
9. subjects who had deep vein thrombosis, myocardial infarction, cerebral infarction or peripheral arterial embolism in the first 12 months
10. Previous history of liver cirrhosis or portal hypertension
11. When screening, alanine aminotransferase, barley transaminase, total bilirubin and blood creatinine are higher than the upper limit of normal value
12. HIV infection or carrier in the past or screening; hepatitis C antibody positive; hepatitis B surface antigen positive or hepatitis B core antibody positive, and HBV-DNA test indicates virus replication
13. Patients with randomized bleeding and/or infection that are still uncontrollable after standardized treatment
14. Uncontrolled hypertension at screening, severe arrhythmia, level III/IV (graded by the New York Heart Association) congestive heart failure
15. Those who are known or suspected to be contraindicated or highly sensitive to Trappa ethanolamine API or cyclosporine
16. The subjects had any malignant solid tumors of the organ system in the first 5 years of screening, regardless of whether they had been treated, metastasis or relapsed, except for local skin basal cell carcinoma; subjects with blood tumors found in the past or screening
17. Pregnant or lactating women
18. Male subjects of women of childbearing age or partners of women of childbearing age refuse to use acceptable contraceptive measures from the period of taking the drug to 28 days after the last time of taking the drug.
19. Randomly participated in other clinical trials and took research drugs in the first 3 months.
20. The researchers believe that there is any situation that may cause the subject to be unable to complete the study or pose an obvious risk to the subject, or other factors that reduce the possibility of joining the group.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Full hematological response rate | About 13 weeks from the first medication to the evaluation.

SECONDARY OUTCOMES:
Partial hematological response rate and total hematological response rate | About 13 weeks from the first medication to the evaluation
Hematological response rate | About 26 weeks from the first medication to the evaluation
The time required for the first hematological response | About 26 weeks from the first medication to the evaluation
Changes in platelet count relative to the baseline of each visiting point of view | About 26 weeks from the first medication to the evaluation
Changes in hemoglobin relative to the baseline of each visiting point of view | About 26 weeks from the first medication to the evaluation
Changes in absolute neutrophil count relative to the baseline of each visiting point of view | About 26 weeks from the first medication to the evaluation
Changes in reticulocyte count relative to the baseline of each visiting point of view | About 26 weeks from the first medication to the evaluation
Cumulative proportion of patients who need blood transfusion | About 26 weeks from the first medication to the evaluation
Cumulative total amount of platelet transfusions | About 26 weeks from the first medication to the evaluation
Cumulative amount of red blood cell infusions | About 26 weeks from the first medication to the evaluation
Cumulative proportion of patients with disease progression | About 26 weeks from the first medication to the evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided